CLINICAL TRIAL: NCT02675192
Title: Biological Aging of Skeletal Muscles in Humans, a Monocentric, Prospective Study
Brief Title: Biological Aging of Skeletal Muscles in Humans
Acronym: BioAge
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ecole Nationale Superieure Lyon (Unknown); Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); Region Rhone Alpes (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1508145; 2015-A01484-45 (Other: ANSM)
Record Dates: First submitted 2016-01-25; First posted 2016-02-05 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-05

CONDITIONS: HEALTHY
Keywords: sarcopenia; elderly; muscle biopsy
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urinary and blood samples will be taken, and a muscle biopsy will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Proof cohort : muscular assessment: * Clinical examination : Body weight, BMI, cardiac frequency, muscular examination,...
  * Blood appraisal : glycaemia, lipidic appraisal, leptin, albumin, coagulation, metabolome and epigenetic tests,...
  * Urinary collection : metabolome tests
  * Maximal voluntary quadriceps strength (MVC)
  * Checking muscle functional skills
  * Muscular biopsy
  Interventions: Other: Proof cohort : muscular assessment

INTERVENTIONS:
Other: Proof cohort : muscular assessment — Clinical examination, blood appraisal, urinary collection, MVC, checking muscle functional skills and muscular biopsy will be performed.

SUMMARY:
Aging affects almost all the tissues and physiological functions, and skeletal muscle is the most affected organ. The progressive decline of the weight and the muscular function linked to the aging contributes to the lack of autonomy and dependence, but also to an increase of the mortality risks. Sarcopenia is also a prevalent condition, because it is detected in 13-24% of 60 years old, and 50% of 80 years old and more.

However, strong inter-individual variations of this prevalence of sarcopenia exists. The key issue is to understand why the biological aging of the skeletal muscle is so different between people.

In this study, mechanisms involved in biological aging of the skeletal muscle in aging people (same chronological age) will be specified.

DETAILED DESCRIPTION:
Aging affects almost all the tissues and physiological functions, and skeletal muscle is the most affected organ. The progressive decline of the weight and the muscular function linked to the aging contributes to the lack of autonomy and dependence, but also to an increase of the mortality risks. Sarcopenia is also a prevalent condition, because it is detected in 13-24% of 60 years old, and 50% of 80 years old and more.

However, strong inter-individual variations of this prevalence of sarcopenia exists. Some elderly (60 years old) reveal a biological aging of 80 years old, whereas 60 years old people reveal a biological aging of 60 years old. The key issue is to understand why the biological aging of the skeletal muscle is so different between people.

Previous sarcopenia studies in Humans did not really focus on chronological aging, they were all based on a comparison between young and old people. No study considered inter-individual modifications (biological aging) in sarcopenia. Furthermore, few studies were associated in the same study to "omic", histological, and epigenetic data, to obtain integrated point of view of Human Sarcopenia.

In this study, mechanisms involved in biological aging of the skeletal muscle in aging people (same chronological age) will be specified.

ELIGIBILITY:
Inclusion Criteria:

* Belonging to the Proof cohort
* Between 80 and 83 years old
* Informed consent signed
* Genetic analyses consent signed
* Subject affiliated or entitled to a social security scheme

Exclusion Criteria:

* Anti coagulative treatment
* Severe obesity (>35)
* All chronic pathology requiring a treatment
* Severe renal insufficiency (discovery less than 6 months)
* Abnormal coagulation appraisal
* Allergy to local anesthetics
* Installation of a prosthetic hip and / or knee in the last six months
* Senile dementia
* Refusal of genetic study

Ages: 80 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients are recruited in the Proof cohort (Barthélemy et al., 2007).
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
The area of type IIA fibers called vastus lateralis. | Day 15
  The primary endpoint is the cross sectional area (measured in µm2) of type IIA fibers from the vastus lateralis muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: FEASSON Léonard, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barthelemy JC, Pichot V, Dauphinot V, Celle S, Laurent B, Garcin A, Maudoux D, Kerleroux J, Lacour JR, Kossovsky M, Gaspoz JM, Roche F. Autonomic nervous system activity and decline as prognostic indicators of cardiovascular and cerebrovascular events: the 'PROOF' Study. Study design and population sample. Associations with sleep-related breathing disorders: the 'SYNAPSE' Study. Neuroepidemiology. 2007;29(1-2):18-28. doi: 10.1159/000108914. PMID 17898520